CLINICAL TRIAL: NCT06576531
Title: Exercise and Prediabetes After Renal Transplantation
Acronym: EXPRED-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Laguna (Other)
Collaborators: Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other)
Responsible Party: Principal Investigator, Raúl Morales Febles, PhD-Physiotherapist, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUC_2022_40
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: PreDiabetes; Kidney Transplantation
Keywords: Adherence; Post-transplant Diabetes Mellitus; Prediabetes; Renal Transplantation; Therapeutic Exercise
MeSH Terms: conditions — Prediabetic State | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): The experimental group will receive an ad hoc designed stepped exercise intervention supported by adherence monitoring.
  Interventions: Other: Therapeutic exercise
- Control group (No Intervention): The control group will follow standard lifestyle recommendations according to clinical practice.

INTERVENTIONS:
Other: Therapeutic exercise — A stepped training intervention designed ad hoc based on a combination of aerobic and strength exercises.
  Arms: Exercise group

SUMMARY:
The present clinical trial, EXPRED-II, is the continuation of EXPRED-I (NCT04489043).

Objective: to evaluate the feasibility of exercise in the reversibility of prediabetes after transplantation, as a first step to prevent Post-Transplant Diabetes Mellitus (PTDM).

Methodology: a total of 50 patients with prediabetes beyond 12 months after transplantation with capacity to perform exercise will be randomized to standard life-style recommendations as per clinical practice (n=25) or to a stepped ad-hoc designed training intervention (n=25). Prediabetes will be diagnosed based on fasting glucose levels and an Oral Glucose Tolerance Test (OGTT). Patients randomized to exercise will start with aerobic exercise training 5 times/week, 30 min/day for 12 months which may be gradually increased to 60 min/day or combined with strength exercise in the last increment in case of prediabetes persistence. The reversibility/persistence/relapse of prediabetes will be measured with fasting glucose and OGTT every 3 months. The study will last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* ≥ 12 months post kidney transplant
* Stable renal function in the last 3-6 months
* Prediabetes (abnormal fasting glucose 100-125 mg/dl and/or glucose intolerance 140-199mg/dl)
* Ability to perform exercise

Exclusion Criteria:

* Infection, cancer, acute cardiovascular disease, advanced kidney disease, pulmonary hypertension and uncontrolled chronic liver disease.
* Inability to understand the protocol
* Severe psychological illness
* PTDM and/or DM prior to transplantation
* Morbid obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Reversibility of pre-diabetes in kidney transplant population through therapeutic exercise | Baseline and every 3 months (up to 12 months)
  There is an exercise programme to test the impact of this treatment on the reversibility of prediabetes. Thus, the persistance of recurrency of prediabetes assessed by an oral glucose tolerance test (OGTT) at intermediate time points (0, 3, 6, 9 and 12 months) will be checked in order to increase the intensity and duration of exercise training.

SECONDARY OUTCOMES:
Compliance | Baseline and every 1.5 months (up to 12 months)
  To ensure compliance, the following measures will be implemented: (a) contact by phone one time per week, (b) individual interview every month and a half to reinforce lifestyle changes and follow all recommended in the exercise prescription; (c) the use of a gadget (xiaomi mi band) to see daily routines of patients and every training prescription; this analyses the time, frequency, burned calories, velocity and distance, among others, to reach the established goal by the physiotherapist.
Analytics | Baseline and every 3 months (up to 12 months)
  To evaluate the improvements in metabolic risk factors profile: obesity, triglycerides, blood pressure and HDL cholesterol.hemogram (hematocrit, haemoglobin, white blood count), biochemist tests: creatinine, HbA1c, total, LDL and HDL cholesterol, triglycerides, uric acid, hepatic enzymes (ASAT, ALAT), levels of immunosuppression, albumin, creatinine, albuminuria, proteinuria in an isolated urinary samples
Anthropometric measures | Baseline and every 3 months (up to 12 months)
  At baseline and at 3, 6, 9, 12 months: weight in kilograms, height in meters, waist circumference, hip circumference, will be measured. Also, BMI Body mass index (BMI): weight in kilograms divided by the square of the height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- University of La Laguna, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided